CLINICAL TRIAL: NCT03930433
Title: The Effect of Nebivolol in Hypertensive Patients With Coronary Arterial Spasm
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Korea University Guro Hospital (Other); Korea University Ansan Hospital (Other); Severance Hospital (Other)
Responsible Party: Principal Investigator, Soon Jun Hong, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NevibololSpasm
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Coronary Vasospasm
Keywords: Nebivolol
MeSH Terms: conditions — Coronary Vasospasm | interventions — Nebivolol; Diltiazem

STUDY DESIGN:
Intervention Model Description: Group 1: Nebivolol group Group 2: Diltiazem group Group 2: Nebivolol + Diltiazem group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nebivolol group (Active Comparator): Oral Nebivolol 5mg / day (2 weeks) -> 10mg / day (10 weeks)
  Interventions: Drug: Nebivolol
- Diltiazem group (Placebo Comparator): Oral Diltiazem 90mg / day (2 weeks) -> 180mg / day (10 weeks)
  Interventions: Drug: Diltiazem
- Nebivolol+Diltiazem group (Placebo Comparator): Oral Nebivolol 2.5mg / day + Oral Diltiazem 45mg / day (2 weeks) -> Oral Nebivolol 5mg / day + Oral Diltiazem 90mg / day (10 weeks)
  Interventions: Drug: Nebivolol+Diltiazem

INTERVENTIONS:
Drug: Nebivolol — Patients are randomly assigned to a ratio of 1: 1: 1, divided into 3 groups.
  Arms: Nebivolol group
Drug: Diltiazem — Patients are randomly assigned to a ratio of 1: 1: 1, divided into 3 groups.
  Arms: Diltiazem group
Drug: Nebivolol+Diltiazem — Patients are randomly assigned to a ratio of 1: 1: 1, divided into 3 groups.
  Arms: Nebivolol+Diltiazem group

SUMMARY:
The correlation between endothelial dysfunction and the risk of coronary heart disease is well known through previous studies. The degradation of the function of nitric oxide acting on the endothelium of blood vessels is mainly explained by reduction of synthesis, loss due to oxidative stress, and decreased sensitivity to vascular dilatation action. In particular, patients with high blood pressure have been known to have impaired vascular endothelial function through animal experiments and several clinical studies, mainly due to increased biomechanical friction in the blood vessels and decreased biological availability of nitric oxide, which in turn causes incongruity in the production of nitric monoxide and changes in normal vascular dilatation. There have also been reports recently that early diagnosis and treatment may improve endothelial dysfunction and prevent the progression of coronary artery disease. However, the reality is that the drugs available in vasospastic angina patients with endothelial dysfunction are very limited. Until recently, beta-blockers were reported to inhibit vascular dilatation of adrenaline stimuli, a drug corresponding to relative contraindications in vasospastic angina patients, with one study reporting that propranolol cannot, but rather exacerbates, vasospastic angina. However, a series of reports on the vascular dilatation of the recently developed third-generation beta-blockers have reinvented the role of beta-blockers in vasospastic angina, especially nebivolol (selective, continuous beta-blockers) is known to act on β-1 adrenaline receptor blockings and endothelium to create vascular dilatation, and also to stimulate β-3 adrenaline receptors to cause nitric oxide generation and antioxidant effects in the endothelium of blood vessels. Therefore, this clinical trial seeks to find whether nebivolol will inhibit vascular contraction in hypertensive patients and will work in angiospastic angina patients.

ELIGIBILITY:
Inclusion Criteria:

* hypertension (stage I-2: Systolic blood pressure 140-179mmHg and diastolic blood pressure 90-109mmHg)
* 20 to 80 years old
* diagnosed with vasospastic angina through coronary angiography and provocation test
* available to outpatient treatment
* voluntarily signed a written consent to participate in the clinical trial

Exclusion Criteria:

1. Previous history of hypersensitivity to beta blockers or calcium channel blockers
2. History of dementia or accompanying psychiatric illness or history of drug abuse
3. Those who participated in other clinical trials within 1 month before screening
4. A person who is unable to perform compliance with the plan and procedures, or who has been judged by the tester to be in a medical condition inappropriate for participation
5. Study subjects who are taking drugs that can affect the study drug efficacy evaluation (ACE inhibitors, angiotensin blockers, beta blockers other than clinical trial drugs, calcium antagonists other than clinical trial drugs, diuretics other than indapamide). These subjects are allowed to participate after a wash-out period of at least 2 weeks
6. Malignant hypertension (with retinal hemorrhage or papilledema) or known moderate or severe retinopathy (retinal hemorrhage within the last 6 months, visual disturbance, retinal microaneurysm)
7. A history of secondary hypertension and all suspected secondary hypertension: coarctation of the aorta, hyperaldosteronism, renal artery stenosis, Cushing's disease, chromatin-positive cell tumor, polycystic kidney disease, etc.
8. Patients with orthostatic hypotension with symptoms
9. Patients with severe heart disease (heart failure New York Heart Association class 3 and 4), recent 6-month ischemic heart disease (angina pectoris, myocardial infarction), percutaneous coronary intervention, or coronary artery bypass surgery)
10. Patients with severe cerebrovascular disease (stroke, cerebral infarction, cerebral hemorrhage within the last 6 months)
11. Patients with anuria or severe renal failure (creatinine clearance <30 mL / min)
12. Severe liver failure or AST or ALT> 3 times the upper limit of normal, biliary obstruction, biliary cirrhosis, cholestasis
13. Gastrointestinal diseases and surgery patients that may affect the absorption, distribution, metabolism, and excretion of drugs, current active gastritis and gastrointestinal / rectal bleeding that the tester considers clinically significant, active inflammatory bowel syndrome within the last 12 months
14. Pregnant and lactating women, those who have a pregnancy plan during the trial and do not agree with the appropriate method of contraception

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Changes in coronary spasm | Baseline to 12 weeks
  The descriptive statistics (mean subject number, standard deviation, median value, minimum value, and maximum value) of changes in the baseline and 12-week outcomes will be presented for each treatment group, and the comparison between the three groups for ANOVA or ANOVA Kruskal-Wallis test. Changes in each group will be analyzed using Paired t-test or Wilcoxon signed rank test. An ANCOVA analysis will be performed when there are more influencing factors.

SECONDARY OUTCOMES:
Changes in Quality of Life | Baseline to 12 weeks
  Changes in Quality of Life based on Seattle Angina Questionnaire
Changes in mean sitting systolic blood pressure and mean sitting diastolic blood pressure | Baseline to 6, 12 weeks
  Changes in mean sitting systolic blood pressure and mean sitting diastolic blood pressure
Percentage of target blood pressure reached | Baseline to 6, 12 weeks
  Percentage of target blood pressure reached from baseline to 6, 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No